CLINICAL TRIAL: NCT05348174
Title: Randomized Controlled Trial of Virtual Reality Assisted Guided Imagery (VRAGI) for Pain Management in Advanced Cancer Patients: Protocol for Efficacy, Feasibility, and Safety in a Home Setting
Brief Title: Randomized Controlled Trial of Virtual Reality Assisted Guided Imagery (VRAGI) for Pain in Advanced Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114598
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cancer Pain; Oncology; Virtual Reality; Depression, Anxiety
MeSH Terms: conditions — Cancer Pain; Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This prospective, 2x2 randomized controlled trial will be conducted with participants from Prisma Health, a tertiary level health care center based in South Carolina, USA. We evaluate the effects of two two-level factors: "Guided imagery" and "VR immersion" and based on the presence and absence of these factors, the study will have 4 arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants, care providers and investigators will be blinded. Randomization will be done via REDCap software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality Assisted Guided Imagery (VRAGI ) (Active Comparator): 20 participants will be randomized to this arm. Participants in this arm will experience the immersive VR guided imagery on VR Head Mounted Displays (Meta Quest 2). They will experience video content and the accompanying guided imagery and nature soundscapes.
  Interventions: Behavioral: Virtual Reality Assisted Guided Imagery (VRAGI)
- Virtual Reality No Guided Imagery or other audio ( VR No GI or other audio) (Sham Comparator): 20 participants will be randomized to this arm. Participants in this arm will experience the immersive VR visual content on VR Head Mounted Displays (Meta Quest 2) but will not experience the accompanying guided imagery narration or nature soundscapes.
  Interventions: Behavioral: Virtual Reality Assisted Guided Imagery (VRAGI)
- Laptop Assisted Guided Imagery (Laptop AGI) (Active Comparator): 20 participants will be randomized to this arm. Participants in this arm will experience the VR content on laptops. They will not receive the VRHMDs. They will experience video content and the accompanying guided imagery and nature soundscapes on a laptop.
  Interventions: Behavioral: Virtual Reality Assisted Guided Imagery (VRAGI)
- Laptop no Guided Imagery or other audio (Laptop no GI or other audio) (Sham Comparator): 20 participants will be randomized to this arm. Participants in this arm will experience the VR content on laptops. They will not receive the VRHMDs. They will experience only the video content on a laptop and will no experience the accompanying guided imagery or nature soundscapes.
  Interventions: Behavioral: Virtual Reality Assisted Guided Imagery (VRAGI)

INTERVENTIONS:
Behavioral: Virtual Reality Assisted Guided Imagery (VRAGI) — The visual landscape consists of a computer-generated immersive virtual world with nature-based imagery (i.e., trees, birds, mountains, water) and accompanying soundscapes with guided imagery.

SUMMARY:
Introduction Patients with advanced cancer often experience high levels of debilitating pain and pain-related psychological distress. Although there is increasing evidence that non-pharmacological strategies are needed to treat their pain, pharmacologic modalities remain the preferred strategy. Guided imagery is a form of focused relaxation that helps create harmony between the mind and body and has been shown to significantly improve cancer pain. This study presents Virtual Reality Assisted Guided Imagery (VRAGI) as an alternative pain treatment modality. The investigators of this study will conduct a randomized control trial to test its efficacy, feasibility, and safety in the home setting, for patients with advanced cancer.

Methods and Analysis The study will recruit 80 participants from Prisma Health, a tertiary level health care center based in Greenville, South Carolina, USA using a stringent set of inclusion and exclusion criteria. The prospective 6-week, 2x2 randomized controlled trial will randomize participants to four groups: (1) VRAGI, (2) Laptop Assisted Guided Imagery (AGI), (3) VR (no guided imagery or other audio), and (4) laptop (no guided imagery or other audio). Participants allocated to VR groups will be trained to use a head-mounted display (HMD) that immerses them in 3D audio-video content. The non-VR group will use a laptop displaying 2D video content. Content includes relaxing natural scenes across three calendar seasons (spring, summer, fall). Investigators will collect measures pre, during, and post intervention including patient reported outcomes (PROs) of pain, anxiety, depression, fatigue. Additionally, investigators will assess the feasibility, acceptability and safety of VRAGI use in a home setting.

Trial Registration Number

#Pro00114598

Strengths and Limitations

* This study uses a novel design that combines the use of immersive Virtual Reality (VR) technology with guided imagery processes to treat chronic pain in advanced cancer patients.
* Investigators propose a reproducible intervention that can be self-administered in a home setting, thus eliminating the need for trained personnel, transportation modalities, or healthcare facilities.
* VR content will be preloaded onto HMDs, thus eliminating the need for access to the internet and decreasing the variability of the intervention.
* Investigators will collect patient reported outcomes (PROs) on pain, anxiety, depression, fatigue, and opioid use, but not continuous user feedback or biofeedback.
* This study focuses on patients < 65 years of age with advanced cancer. This allows the study to focus on a large group of patients but may limit the overall generalizability of the findings.

DETAILED DESCRIPTION:
Objectives

The primary aim of this pilot study is to measure the improvement in pain using virtual reality assisted guided imagery in participants with advanced cancer. The study will utilize a novel approach where participants will be asked to wear a virtual reality head-mounted display presenting immersive virtual reality assisted guided imagery (VRAGI) content in a home setting. In addition to measuring the improvement in pain, this study seeks to: (1) assess the efficacy of immersive VR assisted guided imagery on patient-reported outcomes (PROs), including anxiety and opioid use among patients with advanced cancer (2) measure feasibility, acceptance, and safety of VR-assisted guided imagery in a home setting. The study will recruit 80 participants from Prisma Health Upstate Outpatient Cancer Clinics, who will be randomized to four groups after enrollment:

Participants in all groups will continue to receive the current standard of symptom management treatment. Eligible participants in the VR group will be trained to use a VR head-mounted display (HMD) in the comfort of their own home for self-treatment of cancer pain. The objective is to gather data on participants with advanced cancer after being exposed to 3 weeks of Virtual Reality Assisted Guided Imagery (VRAGI). The study will collect patient reported outcomes (PROs) including pain, anxiety, depression, fatigue, and opioid use. The investigators will also measure feasibility, acceptability and safety of VRAGI at home. The investigators will also collect qualitative data following participants' VR experience to better understand patients' preferences, thoughts, and feelings about the VR experience. Outcomes will be measured before, during, and after a three-week intervention period and compared with the control group. The investigators expect that this study will demonstrate that VRAGI is an effective non-pharmacologic treatment for the management of cancer pain; moreover, the investigators expect VRAGI will be feasibly and safely deployed in home settings.

Study Design Randomized control trial: The study will recruit 80 participants. Once recruited, participants will be screened using the inclusion and exclusion criterion to ensure study eligibility. Eligible participants will be randomized to the intervention and control groups using Redcap software.

Setting The study will recruit 80 participants from Prisma Health Cancer Institute Outpatient Clinics. Once recruited, participants will be screened using the inclusion and exclusion criterion to ensure study eligibility. Participants will experience the intervention in a home setting. Investigators will evaluate the effects of two two-level factors: "Guided imagery" and "VR immersion." The four arms of the study consists of: (1) VRAGI, (2) Laptop AGI, (3) VR (no guided imagery or other audio), and (4) laptop (no guided imagery or other audio). Randomization of participants will be performed via Research Electronic Data Capture (REDCap) using a 1:1:1:1 allocation between the four study groups. During recruitment, we will randomly assign participants who fulfill the inclusion and exclusion criteria to one of the four study groups while balancing age, gender, and cancer progression. Eligible participants in the VRAGI or VR (no GI or other audio) arms will be trained to use a VR head-mounted display (HMD) at home. Participants in the other two groups will use a laptop to watch the same visual content shown in the HMDs. Treatment sessions will last 15-20 min and will occur once a day for three weeks.

Our sample size of 80 is based on an observed mean for pain at baseline of 7 (SD=1, range=0-10), significance level of 0.05, power of 0.8, and anticipated main effect size of 0.6.45 Since recruitment is staggered and the study is completed in batches due to the limited availability of VR headsets, any attrition will be overcome in future waves of recruitment.

Pre-Screening Potential participants will be identified by palliative care and medical oncology providers at the Prisma Health Cancer Institute. Informed consent from participants will be obtained in person by the provider. Participants will have adequate time to ask questions. On receipt of the signed consent form and prior to randomization, participants will be enrolled in a 7-day screening week

Screening Phase The clinical research coordinator will screen consented participants for eligibility using patient electronic health records (EHR) and conduct a phone assessment with potential participants. The study coordinator will screen participants using the inclusion and exclusion criterion. Participants who meet the inclusion criterion will effectively be ruled eligible unless they meet any of the exclusion criteria.

The study coordinator will verify eligibility by a phone call. Eligible participants that do not opt-out will be emailed a recruitment letter and informational brochure. This screening week is designed to evaluate willingness and ability to respond to emailed survey questionnaires, ESAS and Brief Pain Inventory (BPI) forms, which participants are required to respond within the week. The average score of symptoms on ESAS will be used to calculate the baseline (pre-intervention) symptom intensity. A screening failure for this study is defined as a participant who completed fewer than 75% of the forms provided during the screening week. Participants who successfully complete the screening week will be randomized to the 4 study arms. Each arms will recruit 20 patients.

All participants who successfully complete the screening week will receive a second phone call from the study coordinator for an onboarding session. VR HMDs will be mailed out to participants in the VR arms in advance of this call and asked to watch a 10 min video on how to use the HMD. Participants will have unlimited access to these training videos. The study coordinator will discuss the patient packet, which will contain all study instructions and surveys. The study coordinator will be available to support participants throughout the study via phone call and email support. All participants are allowed to undergo any concomitant treatment prescribed by their provider outside of those listed in exclusion criteria.

Intervention Phase The Meta Quest 2 HMD (formerly named Oculus Quest 2) will be used with the VR groups. Participants will be instructed to sit down while viewing VR content. The VRAGI sessions are pre-loaded so that the internet is not needed. Before participants receive their HMD, it will be sanitized via skin friendly antibacterial cleaning wipes and exposing them to ultraviolet light treatment in a CleanBox for one min killing 99.99% of all bacteria including COVID-19 and its variants.

The visual landscape consists of a computer-generated immersive virtual world with nature-based imagery (i.e., trees, birds, mountains, water) and accompanying soundscapes with guided imagery. Participants will complete the sessions in the correct calendar order. The content was developed by an interdisciplinary collaboration of physicians, mental health counselors, human systems engineers, and VR content experts. Participants in all four arms of the study will visually see these virtual worlds. For the two groups containing guided imagery, there will be an accompanied nature-based soundscape (i.e., water flowing, birds chirping, narration). For the two groups containing no guided imagery, there will be no audio provided. Participants are requested to fill out the surveys during the intervention phase, per the study protocol. Surveys will be administered electronically and participants do have the option to complete these on paper as well. Paper surveys will be provided to participants in the patient packet.

Week 1

Pre and Post VR Session (daily):

Complete numerical rating scale for pain, anxiety, depression, fatigue Complete Brief Pain Inventory (Beginning and end of first week) Complete Edmonton Symptom Assessment Scale (Beginning and end of first week) Complete Client Satisfaction Questionnaire (CSQ) (end of first week) Complete VR questionnaire (end of first week) Week 2

Pre and Post VR Session (daily):

Complete numerical rating scale for pain, anxiety, depression, fatigue Complete Brief Pain Inventory (Beginning and end of second week) Complete Edmonton Symptom Assessment Scale (Beginning and end of second week) Complete Client Satisfaction Questionnaire (CSQ) (end of second week) Complete VR questionnaire (end of second week) Week 3

Pre and Post VR Session (daily):

Complete numerical rating scale for pain, anxiety, depression, fatigue Complete Brief Pain Inventory (Beginning and end of third week) Complete Edmonton Symptom Assessment Scale (Beginning and end of third week) Complete Client Satisfaction Questionnaire (CSQ) (end of third week) Complete VR questionnaire (end of third week)

Once the intervention is completed, the participant will mail back the laptops/ HMDs using the prepaid shipping labels provided . Once the laptops and HMDs are received by the research assistant VR-use data will be downloaded from the devices. Before being given to the next set of participants, the HMDs will be cleaned with a CleanBox UV box, which kills 99.9999% of bacteria, viruses, and fungi including SARS-CoV2.

Post-Intervention Phase (Week 6). Complete Brief Pain Inventory (end of week 6). Complete Edmonton Symptom Assessment Scale (end of week 6). At this point the study will be completed for this patient. Participants will continue to follow-up as normal with their physicians at Prisma Health Upstate Outpatient Cancer Clinics.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Advanced cancer, defined as cancer that is incurable including locally advanced and metastatic cancers, with no plan for resection during the study period.
3. Baseline pain score Edmonton Symptom Assessment Scale (ESAS) ≥ 4 (mean score during the screening week).
4. Able to provide consent and willing to comply with all study procedures, as well as comprehend spoken and written English.
5. Have access to a compatible Android, iOS smartphone, personal laptop, or desktop computer (excluding tablets) to complete surveys and respond to emails

Exclusion Criteria:

1. Have a condition that interferes with VR usage including history of seizure, facial injury precluding safe placement of an HMD, or other visual or hearing impairment that impacts ability to participate.
2. Participated in a previous VR clinical study.
3. Underwent a surgical procedure within 8 weeks.
4. Have a neurocognitive disorder according to past medical history.
5. Have brain metastases.
6. Have a prognosis of <3 months from the time of enrollment per treating oncologist.
7. Experience current substance abuse.
8. Experienced complex childhood trauma.
9. Diagnosed with serious mental illness.
10. >65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Chane in Pain score | End of week 1,2, 3 and 6
  Change in pain interference as assessed with the Brief Pain Inventory (BPI) [ Time Frame: Pre-Intervention(baseline), weekly at the end of week 1, 2, 3, and week 6] Pain will be assessed with the Brief Pain Inventory (BPI). Patients will rate their pain from 0=no pain to 10=worst pain imaginable in response to items such as "average pain," "worst pain" and "least pain" over the last 7 days and "pain right now". An average of the responses to these items is used to create a single pain severity score.

SECONDARY OUTCOMES:
Change in Anxiety score, Edmonton Symptom Assessment Scale (ESAS) | end of week 1, 2, 3 and 6
  Change in anxiety score as assessed with the Edmonton Symptom Assessment Scale (ESAS) [ Time Frame: Pre-Intervention(baseline), at the end of week 1, 2, 3 and week 6] Symptoms will be assessed using Edmonton Symptom Assessment Scale (ESAS). Patients will rate their symptoms from 0=no symptom to 10=worst. An average of the responses to these items is used to create a single symptoms severity score .
Change in Depression score, Edmonton Symptom Assessment Scale (ESAS) | end of week 1, 2, 3 and 6
  Change in depression score as assessed with the Edmonton Symptom Assessment Scale (ESAS) [ Time Frame: Pre-Intervention(baseline), at the end of week 1, 2, 3 and week 6] Symptoms will be assessed using Edmonton Symptom Assessment Scale (ESAS). Patients will rate their symptoms from 0=no symptom to 10=worst. An average of the responses to these items is used to create a single symptoms severity score .
Percentage reduction in opioid use | Daily assessed In a 6-week period. Comparing the change from study baseline to Day 7, Day 14, Day 21 and Day 42 in MME of prescribed medication.
  Opioid use will be measured at the start of the study and week 1,2,3 and 6, using an Opioid Diary that will be maintained by the patient.
Proportion of participants that completed intervention per study protocol. | Assessed at the end 6 weeks
  Measured by percentage of patients that adherence to the study protocol. ≥75% of adherence to study protocol is required to determine that the study is feasible.
Proportion of participants that develop adverse events. | Assessed on Day 1 and then weekly at end of week 1, 2 and 3
  Safety of the VR protocol will be assessed based on participants' report of VR side effects. Immediately post intervention, on Days 1, 7, 14 and 21, participants will answer yes or no to a question if they experienced anything uncomfortable, distressing or upsetting as a result of using VR. If yes, the survey allows the participant to describe this.
Median acceptability score. | Assessed weekly at end of week 1, 2, 3 and 6
  Median value from weekly post-intervention survey question asking whether participants would recommend VRAGI to another participant on a scale from 0 (definitely not) to 10 (definitely yes).

CONTACTS AND LOCATIONS:
Overall Officials: Teny Henry Gomez, MD, Principal Investigator — Prisma Health-Upstate
Locations (3):
- United States (3):
  - Clemson University, Clemson, South Carolina
  - Watermark Counseling, Columbia, South Carolina
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No
Data from this study will only be accessible for to the investigators in this team. We do not plan to share IPD with other researchers.

REFERENCES:
- [Background] Birckhead B, Eberlein S, Alvarez G, Gale R, Dupuy T, Makaroff K, Fuller G, Liu X, Yu KS, Black JT, Ishimori M, Venuturupalli S, Tu J, Norris T, Tighiouart M, Ross L, McKelvey K, Vrahas M, Danovitch I, Spiegel B. Home-based virtual reality for chronic pain: protocol for an NIH-supported randomised-controlled trial. BMJ Open. 2021 Jun 15;11(6):e050545. doi: 10.1136/bmjopen-2021-050545. PMID 34130965
- [Background] Zeng Y, Zhang JE, Cheng ASK, Cheng H, Wefel JS. Meta-Analysis of the Efficacy of Virtual Reality-Based Interventions in Cancer-Related Symptom Management. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419871108. doi: 10.1177/1534735419871108. PMID 31441352
- [Background] Banos RM, Espinoza M, Garcia-Palacios A, Cervera JM, Esquerdo G, Barrajon E, Botella C. A positive psychological intervention using virtual reality for patients with advanced cancer in a hospital setting: a pilot study to assess feasibility. Support Care Cancer. 2013 Jan;21(1):263-70. doi: 10.1007/s00520-012-1520-x. Epub 2012 Jun 13. PMID 22688373
- [Derived] Hartshorn G, Browning M, Chalil Madathil K, Mau F, Ranganathan S, Todd A, Bertrand J, Maynard A, McAnirlin O, Sindelar K, Hernandez R, Henry Gomez T. Efficacy of virtual reality assisted guided imagery (VRAGI) in a home setting for pain management in patients with advanced cancer: protocol for a randomised controlled trial. BMJ Open. 2022 Dec 5;12(12):e064363. doi: 10.1136/bmjopen-2022-064363. PMID 36576188